CLINICAL TRIAL: NCT05278988
Title: A Study of Ultrashort PRS Regimen V in the Treatment of MDR-TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Shanghai Public Health Clinical Center (Other Government); No.85 Hospital, Changning, Shanghai, China (Other); Ganzhou Fifth People's Hospital, China (Unknown); Weifang Second People's Hospital, China (Unknown); Anhui Chest Hospital (Other); Fourth Taiyuan People's Hospital, China (Unknown); Shanghai Pudong New Area Pulmonary Hospital, China (Unknown); Huashan Hospital (Other); Zhengzhou Sixth People's Hospital, China (Unknown)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Director, Head of Tuberculosis Department,Shanghai Pulmonary Hospital, Principal Investigator, Clinical Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K21-024
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: MDR-TB
Keywords: MDR-TB; Delamanid; bedaquiline
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Treatment according to WHO MDR-TB treatment guidelines (2019).
  Interventions: Drug: MDR-TB Treatment Regimen(WHO)
- Group B(PRS Regimen V) (Experimental): bedaquiline, delamanid, clofazimine, pyrazinamide
  Interventions: Drug: PRS Regimen V

INTERVENTIONS:
Drug: PRS Regimen V — PRS Regimen V(bedaquiline, delamanid, clofazimine, pyrazinamide)
  Arms: Group B(PRS Regimen V)
Drug: MDR-TB Treatment Regimen(WHO) — Treatment according to WHO MDR-TB treatment guidelines (2019)
  Other Names: WHO Regimen
  Arms: Group A

SUMMARY:
This is an exploratory, prospective, randomized, active control, and open label clinical trial to evaluate the efficacy and safety of 6-9 months treatment with the ultrashort PRS Regimen V.

DETAILED DESCRIPTION:
Shortening the course of treatment based on effective therapy can significantly improve patient compliance and reduce the public health burden.Research on optimal drug combination regimens to further shorten the duration and improve the efficacy of multidrug-resistant tuberculosis treatment is an important research direction.The PRS (parabolic response surface, FSC.II) system is an enhanced use of FSC to better identify and optimize optimal drug combinations.In preliminary studies, it was determined that PRS Regimens V （bedaquiline, delamanid, clofazimine, pyrazinamide）was superior to other regimens and would be a promising combination for XDR-TB because it does not contain fluoroquinolones or aminoglycosides. Preliminary trials have demonstrated that this regimen (PRS Regimens IV) can significantly reduce the duration of treatment required for MDR-TB and achieve a relapse-free cure.

Therefore, the investigators conducted an exploratory, prospective, randomized, positive-controlled, open, multicenter clinical study of this new regimen to observe the efficacy, safety, and recent relapse rate of the new regimen in the treatment of multidrug-resistant tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated newly diagnosed patients with rifampicin resistant (RR) or multidrug resistant (MDR)-TB.
2. Newly treated patients: at least twice confirmed by molecular biology or phenotypic drug susceptibility test to have RR- or MDR-TB; Retreated patients: confirmed once by molecular biology or phenotypic drug susceptibility test to have RR- or MDR-TB.
3. Age between 18 and 65.
4. No abnormality on EKG.
5. Able to understand and sign informed consent form.

Exclusion Criteria:

1. Presence of extrapulmonary TB (including tuberculous pleurisy);
2. History of allergic reaction to any of the drugs used in the study;
3. Presence of any of the following conditions that can lead to prolonged QT:

   1. During screening process, ECG shows QT or QTc interval ≥ 450 ms (permit one non-prescheduled retest within the screening period to re-evaluate the testees' qualification);
   2. Pathological Q waves (any Q wave duration of > 40 ms or depth > 0.4-0.5 mV);
   3. Evidence of ventricular pre-excitation (such as Wolff-Parkinson-White Syndrome);
   4. EKG shows evidence of complete or clinically significant incomplete left or right bundle branch block;
   5. Evidence of 2nd or 3rd degree heart block;
   6. Intraventricular conduction delay, QRS durations > 120 ms;
   7. Slow heart rate, defined as sinus heart rate < 50 bpm;
   8. Having personal or family history of long QT syndrome;
   9. Having heart disease, symptomatic or asymptomatic arrhythmia, excluding sinus arrhythmia;
   10. Fainting (i.e., cardiogenic fainting, not including vasovagal syncope or seizure)
   11. Having risk factors for Torsade de pointes ventricular tachycardia (e.g. heart failure, hypokalemia, hypomagnesemia)
4. Pregnancy or liver, kidney, metabolic, autoimmunity, neurological, psychological or endocrine disease, blood system disease, malignant cancer, long-term users of immunosuppressant drugs.
5. Alcoholism
6. Any patients, based on the judgement of the study medical researchers who are not suitable to participate in the trial or unlikely to complete the trial.
7. Participating in another clinical trial at the same time.
8. History of non-compliance in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
patient cure rate | Through study completion, an average of 18 months
  Assessment of cure rate :
  1. Cure.
  2. Treatment completion.
  3. Treatment failure.
  4. Death.
  5. Loss.
  6. Inconclusive.
  7. Treatment success.

SECONDARY OUTCOMES:
Early bactericidal activity (EBA) | treatment initiation (Day 0; D0) and on Day 2 (D2), Day 7 (D7), and Day 14 (D14) after the start of treatment
  Collect patient sputum between 16:00 to 8:00 the next morning before taking drugs prior to treatment initiation (Day 0; D0) and on Day 2 (D2), Day 7 (D7), and Day 14 (D14) after the start of treatment
Time to culture positivity | Through study completion, an average of 18 months
  culture using MGIT 960 and observe the time to detection of positive growth.
Sputum conversion rate | Through study completion, an average of 18 months
  ompare patient sputum conversion rate between the two groups at one month and two months.
Radiology changes | Through study completion, an average of 18 months
  "Significant absorption" is defined as lesion absorption ≥ ½. "Absorption" is defined as lesion absorption ≤ ½. "No change" if the original lesion has no clear change. "Worsened" if the original lesion is enlarged or has spread. "Closure" if the original cavity is enclosed or enclosed by blockage. "Shrinkage" if diameter of the original cavity decreased by ≥1/2. "No change" if diameter of the original cavity decreases by <1/2. "Enlarged" if diameter of the original cavity increases by >1/2.
Relapse rate one and two years after treatment completion. | At 3, 6, 12, 18, and 24 months
  follow up at 3, 6, 12, 18, and 24 months after treatment completion
Time to Cure by Primary Endpoint criteria | 6-9 month
  Time to Cure by Primary Endpoint criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sha wei, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aung KJ, Van Deun A, Declercq E, Sarker MR, Das PK, Hossain MA, Rieder HL. Successful '9-month Bangladesh regimen' for multidrug-resistant tuberculosis among over 500 consecutive patients. Int J Tuberc Lung Dis. 2014 Oct;18(10):1180-7. doi: 10.5588/ijtld.14.0100. PMID 25216831
- [Background] Van Deun A, Maug AK, Salim MA, Das PK, Sarker MR, Daru P, Rieder HL. Short, highly effective, and inexpensive standardized treatment of multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):684-92. doi: 10.1164/rccm.201001-0077OC. Epub 2010 May 4. PMID 20442432
- [Background] Silva A, Lee BY, Clemens DL, Kee T, Ding X, Ho CM, Horwitz MA. Output-driven feedback system control platform optimizes combinatorial therapy of tuberculosis using a macrophage cell culture model. Proc Natl Acad Sci U S A. 2016 Apr 12;113(15):E2172-9. doi: 10.1073/pnas.1600812113. Epub 2016 Mar 28. PMID 27035987
- See also: WHO consolidated guidelines on drug-resistant tuberculosis treatment — https://apps.who.int/iris/bitstream/handle/10665/311389/9789241550529-eng.pdf?ua=1